CLINICAL TRIAL: NCT07305298
Title: Mirabegron in Patients With Age-Related Macular Degeneration Treated for Overactive Bladder: A Study Protocol for a Non-Randomized Prospective Controlled Trial
Brief Title: Mirabegron in Patients With Age-Related Macular Degeneration
Status: Not yet recruiting | Type: Observational
Sponsor: University of Naples (Other)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Mario Damiano Toro, Principal Investigator, MD, PhD, University of Naples
Other Study IDs: 2025a45673
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Dry AMD; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mirabegron arm: Mirabegron will be administered per os at the dose of 50 mg/day for 12 months
  Interventions: Drug: Mirabegron 50mg
- Control arm: Solifenacin will be administered per os at the dose of 5mg/day for 12 months
  Interventions: Drug: Solifenacin 5mg

INTERVENTIONS:
Drug: Mirabegron 50mg — Mirabegron (50mg/day per os) will be administered in patients with dry AMD and overactive bladder (MMirabegron arm)
  Groups: Mirabegron arm
Drug: Solifenacin 5mg — Solifenacin (5mg/day per os) will be administered in control group (dry amd and overactive bladder)
  Groups: Control arm

SUMMARY:
The goal of this clinical trial is to learn if Mirabegron works to treat dry AMD in patients, aged between 50 and 80 years-old, with early or moderate dry AMD and overactive bladder.

The main question it aims to answer is:

• Is there any change in outer retina morphology in patients treated?

Researchers will compare the safety and efficacy of mirabegron versus conventional approach (Solifenacin) to treat dry AMD in patients with dry AMD and overactive bladder.

Participants will:

* Take Mirabegron or Solifenacin every day for 12 months
* Visit the clinic once every 6 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Age subjects 50 and 80 years-old
* Ability to express informed consent
* Early or moderate dry AMD according to ARDS classification
* Overreactive bladder
* Visual acuity greater than BCVA 65 EDTRS letters.

Exclusion Criteria:

* • Any medical condition which contraindicates the use of beta-agonists

  * Uncontrolled hypertension
  * Tachycardia or atrial fibrillation
  * Any allergies to the beta-agonists
  * Renal or hepatic failure
  * Long QT or concomitant treatment with drugs that cause lengthening of the QT interval
  * Any sign of ocular inflammation
  * xudative AMD
  * Any ongoing medical or surgical treatment for AMD (including intravitreal injections, oral supplementation of lutein, zeaxanthin and or high dietary intake of antioxidants)
  * Any other ophthalmic diseases such glaucoma, acute or chronic uveitis, advanced cataract, or any opacities of the ocular media that do not permit high-quality imaging examinations.
  * Pregnancy
  * Any condition or disease that in the opinion of the investigators may put the subject at significant risk or may interfere significantly with the subject's participation in the study (i. e. malignancy, uncontrolled or cardiovascular diseases)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects aged between 50 and 80 years-old with early or moderate dry AMD and overreactive bladder treated with either Mirabegron or Solifenacin
Sampling Method: Non-Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in outer retinal morphology using SD-OCT | "From enrollment to the end of treatment at 12 months
  Outer nuclear layer (ONL) thickness, choroidal thickness (ChT), central macular thickness (CMT) will all be measured in micron
Changes in FAF assessing | "From enrollment to the end of treatment at 12 months
  changes in FAF measured in micron

SECONDARY OUTCOMES:
mean BCVA | From enrollment to the end of treatment at 12 months
  Mean BCVA according to the ETDRS charts
Mean macular sensitivity (MS) | From enrollment to the end of treatment at 12 months

OTHER OUTCOMES:
Safety parameters | From enrollment to the end of treatment at 12 months
  blood pressure measured in mmHg
Safety parameters | From enrollment to the end of treatment at 12 months
  heart frequency in bpm
Safety parameters | From enrollment to the end of treatment at 12 months
  SpO2 (Peripheral Oxygen Saturation) in % saturation
Safety parameters | From enrollment to the end of treatment at 12 months
  Respiratory rate in dpm

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II, Naples, Italy